CLINICAL TRIAL: NCT00942136
Title: The Official Study Title Exceeds the 300 Character Limit for This Field. See Detailed Study Description Section for Official Study Title.
Brief Title: GSK1349572 Proton Pump Inhibitor Drug Interaction and Supratherapeutic Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112941
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Healthy Volunteer
Keywords: HIV; GSK1349572; omeprazole; Prilosec; supratherapeutic dose; pharmacokinetics; drug interaction; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Omeprazole

ARMS (3):
- Cohort 1, Sequence 1 (Experimental): Subjects in Cohort 1, Sequence 1 will receive a single dose of GSK134972 50 mg after a fast of 10 hours in Period 1. Following a 7 day washout, they will receive a single dose of GSK134972 50 mg after a high fat meal in Period 2. After the last PK sample is collected in Period 2, they will receive a single daily dose of omeprazole 40 mg for 5 days. On Day 5 they will receive a single dose of GSK134972 50 mg 2 hours after the omeprazole dose. Subjects will have a screening visit 30 days prior to the first dose and a follow-up visit 7-14 days after the last dose of medication.
  Interventions: Drug: GSK1349572; Drug: Omeprazole
- Cohort 2 (Experimental): Subjects will receive a single dose of either GSK1349572 250 mg or placebo as a suspension. Subjects will have a screening visit within 30 days prior to the dose of study medication and a follow up visit 7-14 days after the dose of study medication.
  Interventions: Drug: GSK1349572; Drug: Placebo
- Cohort 1, Sequence 2 (Experimental): Subjects in Cohort 1, Sequence 2 will receive a single dose of GSK134972 50 mg after a a high fat meal in Period 1. Following a 7 day washout, they will receive a single dose of GSK134972 50 mg after fast of 10 hours in Period 2. After the last PK sample is collected in Period 2, they will receive a single daily dose of omeprazole 40 mg for 5 days. On Day 5 they will receive a single dose of GSK134972 50 mg 2 hours after the omeprazole dose. Subjects will have a screening visit 30 days prior to the first dose and a follow-up visit 7-14 days after the last dose of medication.
  Interventions: Drug: GSK1349572; Drug: Omeprazole

INTERVENTIONS:
Drug: GSK1349572 — GSK1349572 250 mg suspension as a single dose. GSK1349572 is an investigational (not approved by the FDA) medication for the treatment of HIV in the class of integrase inhibitors.
  Arms: Cohort 2
Drug: GSK1349572 — GSK1349572 50 mg tablets as a single dose on three separate occasions. GSK1349572 is an investigational (not approved by the FDA) medication for the treatment of HIV in the class of integrase inhibitors.
  Arms: Cohort 1, Sequence 1; Cohort 1, Sequence 2
Drug: Placebo — Placebo Suspension as a single dose.
  Arms: Cohort 2
Drug: Omeprazole — Omeprazole 40 mg once a day for 5 days. Omeprazole is approved by the FDA currently to reduce stomach acid, treat stomach ulcers, and gastroesophageal reflux disease.
  Other Names: PRILOSEC. PRILOSEC is a registered trademark of AstraZeneca, LP.
  Arms: Cohort 1, Sequence 1; Cohort 1, Sequence 2

SUMMARY:
GSK1349572 is an integrase inhibitor that is currently being evaluated for the treatment of HIV infection. The primary objective of this study is to determine whether the addition of a proton pump inhibitor, omeprazole, to GSK1349572 impacts the blood levels of GSK1349572. It will also evaluate if a high fat meal impacts the blood levels of GSK1349572. In addition, the safety, tolerability, and pharmacokinetics of single supratherapeutic (high) dose of GSK1349572 will be evaluated.

DETAILED DESCRIPTION:
Official Study Title: A randomized, double-blind study to evaluate the safety, tolerability, and pharmacokinetics of a supratherapeutic dose of GSK1349572 250 mg and a randomized, open-label study to evaluate the effects of omeprazole 40 mg daily and a high fat meal on the pharmacokinetics of GSK1349572 50 mg in healthy adult subjects (ING112941)

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age, inclusive.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory] or, Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 3 days after the last dose of study drug.
* Body weight ≥ 50 kg for men and ≥ 45 kg for women and BMI within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* History of regular use of tobacco or nicotine-containing products within 3 months prior to screening.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* History of sensitivity to any of the study medications, or components thereof including sulfa-containing drugs, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine human hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of significant renal or hepatic diseases.
* History/evidence of clinically significant pulmonary disease.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, inflammatory bowel disease, or pancreatitis should be excluded. Subjects with gastroesophageal reflux disease requiring the use of proton pump inhibitors or H2-blockers.
* History of upper gastrointestinal bleeding.
* Active peptic ulcer disease.
* Subjects with a hemoglobin <12 g/dL. A single repeat is allowed for eligibility determination.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects. A single repeat is allowed to determine subject eligibility.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination) outside of the protocol limits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Plasma GSK1349572 PK parameters following a single-dose administration of 50 mg under fasted conditions with and without omeprazole 40 mg | 16 days
Plasma GSK1349572 PK parameters following a single-dose administration of 50 mg under fasted conditions and with a high-fat meal | 9 days
Plasma GSK1349572 PK parameters following a single-dose administration of 250 mg under fasted conditions | 3 days
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, ECG, and vital signs assessments following a single supratherapeutic dose of GSK1349572 250 mg. | 3 days

SECONDARY OUTCOMES:
Safety and tolerability parameters, including adverse event, concurrent medication, clinical laboratory, ECG, and vital signs assessments following a single-dose administration of 50 mg under fasted conditions, with a high-fat meal, and with OMP 40 mg. | 16 days
Plasma GSK1349572 PK parameters following a single-dose administration of 50 mg under fasted conditions, with a high-fat meal, and with OMP 40 mg | 16 days
Plasma GSK1349572 PK parameters following a single-dose administration of 250 mg under fasted conditions | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States